CLINICAL TRIAL: NCT05193032
Title: Abces After Incision: Recurrence or Not?
Acronym: ABCINCIS
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ABCINCIS
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Anal Abscess; Perianal Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The French School of Proctology assumes that any anal or perianal abscess is related to an anal fistula and therefore requires treatment at the risk of recurrence of the abscess. The Anglo-Saxons, on the other hand, recommend a simple incision in case of a first abscess, without taking care of the possible fistula, on the grounds that more than 60% of patients will not have a recurrence of their abscess. In addition, predictive factors of abscess recurrence have been reported such as female gender, age over 40 years, however, contradicted by other studies. High BMI, corticosteroid use, Crohn's disease are other predictive factors of recurrence while diabetes mellitus or antibiotic therapy during the days following the incision were considered as "protective". The objective of this study was to evaluate our experience in the hospital with essentially a description of the evolution of the patients in the 2 years following the incision of the abscess in consultation.

The main objective is to describe the evolution of patients, within 2 years, who consulted our center for an anal or perianal abscess treated by a simple skin incision under local anesthesia in consultation and/or whose fistula was not found during the examination under anesthesia in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient who visited between January 1, 2019 and December 31, 2019 for an anal or perianal abscess
* Patient who had a skin incision of a first anal margin or buttock abscess and/or whose fistula was not found during examination under anesthesia in the operating room
* French speaking patient

Exclusion Criteria:

* Patient with pilonidal abscess
* Patient with an intramural abscess
* Patient with a history of anal margin or buttock abscess and/or anal fistula
* Patient with a history of proctologic surgery
* Patient with an abscess whose skin incision under local anesthesia has failed
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his or her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients managed at the center for anal or perianal abscesses treated with a simple skin incision under local anesthesia in consultation and/or whose fistula was not found during examination under anesthesia in the operating room, between January 1, 2019 and December 31, 2019
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Evolution of the patients, within 2 years | Year 2
  This outcome corresponds to the rate of occurrence of at least one new abscess, within 2 years, in patients who were treated by a simple skin incision in consultation and/or whose fistula was not found during examination under anesthesia in the operating room.

SECONDARY OUTCOMES:
Predictive factors for recurrence of abscesses | Year 2
  This outcome corresponds to the Predictive factors for the occurrence of at least one new abscess, within 2 years, in patients who consulted our center for an anal or perianal abscess treated by a simple skin incision in consultation and/or whose fistula was not found during the examination under anesthesia in the operating room.
Patient care | Year 2
  This outcome corresponds to the Description of the management (imaging, surgical techniques, number of surgical procedures) of patients who were operated on under anesthesia in the operating room and whose fistula was found.
Cure rate | Year 2
  This outcome corresponds to the Healing and anal incontinence rates of patients who were operated on under anesthesia in the operating room and whose fistula was found.

CONTACTS AND LOCATIONS:
Overall Officials: Amine ALAM, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Quah HM, Tang CL, Eu KW, Chan SY, Samuel M. Meta-analysis of randomized clinical trials comparing drainage alone vs primary sphincter-cutting procedures for anorectal abscess-fistula. Int J Colorectal Dis. 2006 Sep;21(6):602-9. doi: 10.1007/s00384-005-0060-y. Epub 2005 Nov 30. PMID 16317550
- [Background] Malik AI, Nelson RL, Tou S. Incision and drainage of perianal abscess with or without treatment of anal fistula. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD006827. doi: 10.1002/14651858.CD006827.pub2. PMID 20614450
- [Background] Sahnan K, Askari A, Adegbola SO, Tozer PJ, Phillips RKS, Hart A, Faiz OD. Natural history of anorectal sepsis. Br J Surg. 2017 Dec;104(13):1857-1865. doi: 10.1002/bjs.10614. Epub 2017 Aug 31. PMID 28857130
- [Background] Sahnan K, Askari A, Adegbola SO, Warusavitarne J, Lung PFC, Hart A, Faiz O, Phillips RKS, Tozer P. Persistent Fistula After Anorectal Abscess Drainage: Local Experience of 11 Years. Dis Colon Rectum. 2019 Mar;62(3):327-332. doi: 10.1097/DCR.0000000000001271. PMID 30451763
- [Background] Sho S, Dawes AJ, Chen FC, Russell MM, Kwaan MR. Operative Incision and Drainage for Perirectal Abscesses: What Are Risk Factors for Prolonged Length of Stay, Reoperation, and Readmission? Dis Colon Rectum. 2020 Aug;63(8):1127-1133. doi: 10.1097/DCR.0000000000001653. PMID 32251145
- [Background] Lohsiriwat V, Yodying H, Lohsiriwat D. Incidence and factors influencing the development of fistula-in-ano after incision and drainage of perianal abscesses. J Med Assoc Thai. 2010 Jan;93(1):61-5. PMID 20196412
- [Background] He Z, Du J, Wu K, Chen J, Wu B, Yang J, Xu Z, Fu Z, Pan L, Wen K, Wang X. Formation rate of secondary anal fistula after incision and drainage of perianal Sepsis and analysis of risk factors. BMC Surg. 2020 May 6;20(1):94. doi: 10.1186/s12893-020-00762-3. PMID 32375721
- [Background] Mocanu V, Dang JT, Ladak F, Tian C, Wang H, Birch DW, Karmali S. Antibiotic use in prevention of anal fistulas following incision and drainage of anorectal abscesses: A systematic review and meta-analysis. Am J Surg. 2019 May;217(5):910-917. doi: 10.1016/j.amjsurg.2019.01.015. Epub 2019 Jan 31. PMID 30773213